CLINICAL TRIAL: NCT04652297
Title: A Phase I, Randomized, Double-blind, Placebo-controlled Dose Escalation Trial to Assess the Safety Tolerability and Pharmacokinetics of Single and Multiple Oral Administration of HS-10356 in Healthy Volunteers
Brief Title: Safety, Tolerability and Pharmacokinetics of Single and Multiple Oral Administration of HS-10356 in Healthy Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: HS-10356-101
Record Dates: First submitted 2020-11-16; First posted 2020-12-03 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-11

CONDITIONS: Healthy
Keywords: HS-10356; Safety; Pharmacokinetics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HS-10356 single dose (Experimental): Single oral dose of HS-10356 ascending dose
  Interventions: Drug: HS-10356
- placebo single dose (Placebo Comparator): Single oral dose of placebo ascending doses
  Interventions: Drug: Placebo
- HS-10356 multiple doses (Experimental): Multiple oral doses of HS-10356 ascending doses
  Interventions: Drug: HS-10356
- Placebo multiple doses (Placebo Comparator): Multiple oral doses of placebo ascending doses
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HS-10356 — Single dose of HS-10356
  Arms: HS-10356 single dose
Drug: Placebo — Single dose of Placebo
  Arms: placebo single dose
Drug: HS-10356 — Multiple doses of HS-10356
  Arms: HS-10356 multiple doses
Drug: Placebo — Multiple doses of Placebo
  Arms: Placebo multiple doses

SUMMARY:
The primary objective of this study is to assess the safety and tolerability of single and multiple oral administration of HS-10356 in healthy volunteers.

DETAILED DESCRIPTION:
This is a phase I, randomized, double-blind, placebo-controlled, single ascending dose (SAD) and multiple ascending dose (MAD) clinical trial to assess the safety, tolerability, and pharmacokinetics of HS-10356 oral formulation in Chinese healthy adult volunteers.

Approximately five sequential dose panels (single oral doses of 2,6,15,30,45mg HS-10356) will be evaluated in SAD. To protect the safety of volunteers, two sentinel volunteers were first enrolled in the first dose panel (2mg panel) and randomly assigned to HS-10356 or placebo in a 1:1 ratio. After the sentinel volunteers were given the dose for at least 24 hours and confirmed that they were safe, the remaining 6 volunteers were randomly assigned to HS-10356 or placebo in a ratio of 5:1. For the follow-up panels of SAD, volunteers were randomly assigned to either the experimental group or the placebo group (6 cases in HS-10356 and 2 cases in placebo) in a 3:1 ratio using block randomization method. Approximately three sequential dose panels (14 consecutive days for respectively daily oral doses of 6,15,30mg HS-10356, QD) will be evaluated in MAD. Volunteers were randomly assigned to either the experimental group or the placebo group (9 cases in the HS-10356 and 3 cases in the placebo) in a ratio of 3:1 using block randomization method. Each subject will receive only one regimen in this study. Safety data up to Day12 (±2) in SAD and up to Day25 (±2) in MAD will be reviewed prior to dose escalation. Cohorts of SAD and MAD will be added or removed depending on the assessment results of SRC.

ELIGIBILITY:
Inclusion Criteria：

Volunteers must meet all of the following inclusion criteria to be eligible for participation in this study:

1. Full understanding of the content, process and possible adverse reactions of the study, and sign the ICF voluntarily;
2. Healthy Volunteers between 18 and 55 years of age (including the critical value);
3. Male weight is not less than 50 kg, female weight is not less than 45 kg. The body mass index (BMI = weight (kg)/height (m2). The BMI should be controlled within the range of 18 to 26 (including the critical value);
4. Volunteers agree to refrain from smoking, drinking alcohol. Avoid xanthine or caffeine (including chocolate, tea, coffee, cola, etc.) and avoid strenuous exercise;
5. Agreed to use effective contraception from the date of signing of the ICF until six months after the last administration;
6. The male volunteers agreed to refrain from donating sperm from the start of the drug until six months after they stopped the study;
7. The female volunteers agreed to avoid ovum donation from the start of the drug until six months after they stopped the study;
8. Pregnancy test results of female volunteers must be negative within 3 days of administration.

Exclusion Criteria:

1. Pregnant and breastfeeding female.
2. Volunteers with a history of cardiovascular, respiratory, liver, kidney, digestive tract, mental, neurological, hematological, metabolic and other systemic diseases, who are not suitable to participate in this study as assessed by the investigator.
3. The results of vital signs, physical examination, laboratory examination and 12-lead ECG during screening were abnormal with clinical significance.
4. Major surgery was performed within 3 months prior to the screening or surgery was planned during the study.
5. Severe infections, such as cellulitis, pneumonia, sepsis, have occurred or are present in the 30 days prior to screening.
6. ALT, AST, ALP or bilirubin were higher than the upper limit of normal.
7. Creatinine clearance < 90mL/min at screening (Cockcroft-Gault method), as follows:

(140-age in years)×weight (kg)/72×serum creatinine（mg/dL）×(Female×0.85)；

8.Hepatitis B virus surface antigen (HBsAg), hepatitis C virus antibody (HCVAb), human immunodeficiency virus antibody (HIVAb) or syphilis antibody is positive.

9.Volunteers had a history of drug dependence or abuse.

10.A heavy smoker or smokers who smoked 5 or more cigarettes per day for 3 months prior to screening or tested positive for nicotine during screening.

11.A history of alcohol abuse or a single consumption of more than 14 units of alcohol (1 unit = 285 mL of beer, 25 mL of spirits, 150 mL of wine) in the nearly two weeks prior to screening or a positive breath test for alcohol at screening.

12.Participate in clinical trials of any drug or medical device within 3 months prior to screening.

13.Blood donation or blood loss ≥ 400mL within 3 months prior to screening, or blood transfusion received; Blood donation or blood loss ≥ 200mL within 1 month before screening.

14.Volunteers received systemic steroid, immunomodulator, or chemotherapy in the 3 months prior to screening，or likely to be treated with these drugs such as corticosteroids, immunoglobulin, and other immune or cytokine therapy during the study period.

15.Gastrointestinal ulcer, gastroesophageal reflux disease, or other severe symptoms of excess gastric acid secretion.

16.Medical or surgical treatment that permanently alters oral drug absorption and excretion, such as Gastric or intestinal surgery. Cholecystectomy, appendectomy and hernia repair are excluded.

17.Potent CYP3A4 inhibitors and potent CYP3A4 inducers was used within 28 days before administration.

18.Any medication taken within 2 weeks of administration, including prescription, over-the-counter, and herbal medicines.

19.Grapefruit juice, grapefruit and Seville orange juice were consumed in the 2 weeks prior to administration.

20.Diet or dietary treatment or significant change in dietary habits within 30 days prior to administration for whatever reason.

21.Volunteers who have difficulty swallowing solid tablets or capsule. 22.Volunteers with difficulty in blood collection, unable to tolerate multiple venous blood collection and any blood collection contraindications.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Estimated)
Dates: Start 2020-12 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
The incidence, severity, and association of AE, SAE, and adverse events leading to withdrawal from the trial | SAD: Day1~Day12
The incidence, severity, and association of AE, SAE, and adverse events leading to withdrawal from the trial | MAD: Day1~Day25
Laboratory assessment:Haematology | Predose, day 6 prior to discharge from hospital in SAD.
Laboratory assessment:Haematology | Predose, day4、day7、day10、day14、day19 prior to discharge from hospital in MAD
Laboratory assessment:Clinical Chemistry | Predose, day 6 prior to discharge from hospital in SAD.
Laboratory assessment:Clinical Chemistry | Predose, day4、day7、day10、day14、day19 prior to discharge from hospital in MAD
Laboratory assessment:Routine Urinalysis | Predose, day 6 prior to discharge from hospital in SAD.
Laboratory assessment:Routine Urinalysis | Predose, day4、day7、day10、day14、day19 prior to discharge from hospital in MAD
Laboratory assessment:Coagulation test | Predose, day 6 prior to discharge from hospital in SAD.
Laboratory assessment:Coagulation test | Predose, day4、day7、day10、day14、day19 prior to discharge from hospital in MAD
Vital signs:Blood pressure | Within 1 hour before administration,1hour, 2hours, 4hours, 12hours, 24hours, 48hours, 72hours, 96hours, and 120hours after administration in SAD.
Vital signs:Blood pressure | Within 1 hour before administration, 1hours, 2hours, 4hours, 12hours on days 1,2,4,6,8,10,12 and 14, once a day on days 15 to 19 in MAD
Vital signs:Pulse rate | Within 1 hour before administration, 1hour, 2hours, 4hours, 12hours, 24hours, 48hours, 72hours, 96hours, and 120hours after administration in SAD.
Vital signs:Pulse rate | Within 1 hour before administration, 1hours, 2hours, 4hours, 12hours on days 1,2,4,6,8,10,12 and 14, once a day on days 15 to 19 in MAD
Vital signs:Respiratory rate | Within 1 hour before administration, 1hour, 2hours, 4hours, 12hours, 24hours, 48hours, 72hours, 96hours, and 120hours after administration in SAD.
Vital signs:Respiratory rate | Within 1 hour before administration, 1hours, 2hours, 4hours, 12hours on days 1,2,4,6,8,10,12 and 14, once a day on days 15 to 19 in MAD
Vital signs:Temperature | Within 1 hour before administration,1hour, 2hours, 4hours, 12hours, 24hours, 48hours, 72hours, 96hours, and 120hours after administration in SAD.
Vital signs:Temperature | Within 1 hour before administration, 1hours, 2hours, 4hours, 12hours on days 1,2,4,6,8,10,12 and 14,once a day on days 15 to 19 in MAD
Physical examination:General | 2hours, 24hours and 120hours after administration in SAD.
Physical examination:General | 24hours after the first and last administration, prior to discharge from hospital in MAD
Physical examination:Lymph node | 2hours, 24hours and 120hours after administration in SAD.
Physical examination:Lymph node | 24hours after the first and last administration, prior to discharge from hospital in MAD
Physical examination:Chest | 2hours, 24hours and 120hours after administration in SAD.
Physical examination:Chest | 24hours after the first and last administration, prior to discharge from hospital in MAD
Physical examination:Abdominal | 2hours, 24hours and 120hours after administration in SAD.
Physical examination:Abdominal | 24hours after the first and last administration, prior to discharge from hospital in MAD
12-lead electrocardiogram (ECG) parameters ( Heart rate, PR, R-R, QRS and QTcF (average)) | Within 1 hour before administration,1hours, 2hours, 3hours, 24hours 120hours after administration in SAD.

SECONDARY OUTCOMES:
SAD pharmacokinetic endpoint:The maximum plasma concentration (Cmax) | Day1-Day6
SAD pharmacokinetic endpoint:Time to Cmax (Tmax) | Day1-Day6
SAD pharmacokinetic endpoint:The area under the plasma concentration-time curve from time zero to the time of the last measurable concentration (AUC0-t) | Day1-Day6
SAD pharmacokinetic endpoint:The area under the plasma concentration-time curve from time zero extrapolated to infinite time (AUC0-∞) | Day1-Day6
SAD pharmacokinetic endpoint:Terminal rate constant (λz) | Day1-Day6
SAD pharmacokinetic endpoint:Half life (t½) | Day1-Day6
SAD pharmacokinetic endpoint:Apparent clearance following extravascular administration (CL/F) | Day1-Day6
SAD pharmacokinetic endpoint:Apparent volume of distribution following extravascular administration (Vd/F) | Day1-Day6
SAD pharmacokinetic endpoint:Mean residence time (MRT) | Day1-Day6
MAD pharmacokinetic endpoint:The maximum steady state drug concentration in plasma during dosing interval (Css,max) | Day1-Day19
MAD pharmacokinetic endpoint:The minimum steady state drug concentration in plasma during dosing interval (Css,min) | Day1-Day19
MAD pharmacokinetic endpoint:Average steady state drug concentration in plasma during dosing interval (Css,av) | Day1-Day19
MAD pharmacokinetic endpoint:Time to Css, max (Tss,max) | Day1-Day19
MAD pharmacokinetic endpoint:The area under the plasma concentration-time curve over the dosing interval at steady state (AUCss) | Day1-Day19
MAD pharmacokinetic endpoint:The area under the plasma concentration-time curve from time zero to the time of the last measurable concentration at steady state(AUC0-t) | Day1-Day19
MAD pharmacokinetic endpoint:The area under the plasma concentration-time curve from time zero extrapolated to infinite time (AUC0-∞) at steady state | Day1-Day19
MAD pharmacokinetic endpoint:Half life (t½) | Day1-Day19
MAD pharmacokinetic endpoint:Accumulation ratio (Rac) | Day1-Day19
MAD pharmacokinetic endpoint:Apparent clearance at steady state following extravascular administration (CLss/F) | Day1-Day19
MAD pharmacokinetic endpoint:Apparent volume of distribution at steady state following extravascular administration (Vd/F) | Day1-Day19

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China